CLINICAL TRIAL: NCT04306367
Title: A Phase II, Single-arm Study of Combination Pembrolizumab and Olaparib in the Treatment of Patients With Advanced Cholangiocarcinoma
Brief Title: Study of Pembrolizumab and Olaparib in Bile Duct Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000908
Record Dates: First submitted 2020-02-11; First posted 2020-03-12 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — pembrolizumab; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental (Experimental): Pembrolizumab Q3W, IV infusion (day 1 of each 3 week cycle)
  Olaparib bid, Oral tablet continuously
  Interventions: Drug: Pembrolizumab; Drug: Olaparib

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg given intravenously.
  Other Names: Keytruda
Drug: Olaparib — 300 mg given orally.
  Other Names: LYNPARZA

SUMMARY:
The investigators propose an open label, one-arm study to assess the safety and efficacy of olaparib and pembrolizumab in patients with cholangiocarcinoma who have progressed on or cannot tolerate gemcitabine-based therapy.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the ORR of patients with advanced cholangiocarcinoma receiving a combination of pembrolizumab and olaparib. It is hypothesized that the addition of olaparib will improve the response rate of second line systemic therapy from 17.5% to 35% in patients with advanced cholangiocarcinoma.

The study is designed to enroll 33 subjects (for 85% power) with advanced stage cholangiocarcinoma to test the hypothesis that the combination of olaparib and pembrolizumab will increase the ORR in comparison with the ORR from second line systemic chemotherapy (historical control) in this patient population. As the primary study endpoint, which is also being used to determine the sample size of the study, the investigators propose that the combination of olaparib and pembrolizumab will increase the ORR to 35% from 17.5% (achieved with systemic cytotoxic chemotherapy including mFOLFOX-historical control). To allow a 10% patient drop off rate, the investigators expect to enroll a total of 36 subjects into this study. In addition, as secondary study endpoints the investigators expect to see an increase in the PFS and OS of patients receiving combination therapy compared to cytotoxic chemotherapy.

In this study, the investigators propose the collection of three biopsies-one at baseline prior to the start of treatment, one at the beginning of week 4, three weeks after the administration of combination olaparib and pembrolizumab, and one at the time of cancer progression-for the elucidation of exploratory study endpoints. Patients will have a CT or MRI scan at the beginning of treatment and then every 6 weeks thereafter for the first six months of study treatment administration, then every 9 weeks for up to 12 months after the start of treatment, followed by every 12 weeks up to 24 months on study. All patients will continue to receive olaparib and pembrolizumab combination treatment as tolerated unless unacceptable toxicities or cancer progression occur, at which time therapy will cease. In the absence of any problems, the planned study duration is 20-36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be ≥ 18 years of age on day of signing informed consent.
3. Patients must have received 1 line of prior systemic therapy for metastatic or resectable disease (i.e. patients may have received adjuvant gemcitabine and then later platin-based therapy for recurrent metastatic disease)
4. Histological confirmation of cholangiocarcinoma manifesting as either intrahepatic, extrahepatic or gallbladder cancer. Patients with ampullary cancer are excluded.
5. Have measurable disease based on RECIST 1.1.
6. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the sponsor-investigator. Subjects from whom a biopsy is not medically possible or safe may be enrolled on the study upon agreement from the principal investigator.
7. Have a performance status of 0 or 1 on the ECOG Performance Scale.
8. Demonstrate adequate organ function as defined in Table 1. All screening labs will be performed within 28 days of registration.

   Table 1: Adequate Organ Function Laboratory Values System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥ 1,500 /μL Platelets ≥ 100,000 / μL Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment) Renal Serum creatinine OR Measured or calculateda creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤ 1.5 X upper limit of normal (ULN) OR

   ≥ 50 mL/min for subject with creatinine levels > 1.5 x institutional ULN Hepatic Serum total bilirubin ≤ 2.0 X ULN AST (SGOT) and ALT (SGPT) ≤ 3.0 X ULN OR

   ≤ 5 X ULN for subjects with liver metastases Albumin > 2.5 mg/dL Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT)

   Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

   ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants aCreatinine clearance should be calculated per institutional standard.
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section in Appendix 3). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
11. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. A history of anaphylaxis to olaparib
2. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
3. A woman of childbearing potential (WOCBP) who has a positive urine pregnancy test within 72 hours prior to 1st dose of treatment (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
4. Has a known history of active TB (Bacillus Tuberculosis).
5. Has known hypersensitivity to pembrolizumab or any of its excipients.
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   NOTE: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

   NOTE: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has known history of, or any evidence of active, non-infectious pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the site investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
17. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
18. Has known active Hepatitis B without HBV treatment (HBV infection with ongoing HBV treatment is allowed); chronic Hepatitis C infection is allowed. Any patient receiving treatment for HCV should wait at least 14 days after completion of HCV treatment before beginning study treatment. No patient should receive HCV treatment while receiving study treatment. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
19. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-07-16 (Actual); Study Completion 2024-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Marshall, MD, Principal Investigator — Georgetown University
Locations (1):
- Lombardi Comprehensive Cancer Center, Georgetown University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Sadagopan N, Wang H, Yin C, Weinberg BA, Noel MS, Mukherji R, Geng X, Marshall JL, He AR. A phase II single-arm study of combination pembrolizumab and olaparib in the treatment of patients with advanced biliary tract cancer. NPJ Precis Oncol. 2025 Jul 8;9(1):229. doi: 10.1038/s41698-025-01009-1. PMID 40629097

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Pembrolizumab Q3W, IV infusion (day 1 of each 3 week cycle)
  Olaparib bid, Oral tablet continuously
  Pembrolizumab: 200 mg given intravenously.
  Olaparib: 300 mg given orally.
Period: Overall Study
Arm/Group | Experimental
Started | 14
Completed | 1
Not Completed | 13
Not completed — Progression of Disease | 9
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The objective response rate (ORR) is the number of subjects with confirmed Partial Response or Complete Response according to RECIST 1.1, for target lesions assessed by Computed tomography (CT) Scan.
Time Frame: up to 2 years
Population: 1 subject only received 1 cycle, so was not included in ORR.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 13
Participants | 2

2. Secondary Outcome: Duration of Response
Description: Duration of response (DOR), number of months from first response to progression.
Time Frame: 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Experimental
Number analyzed (Participants) | 13
months | 19.75 [6.1 to 33.4]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) is the time from enrollment to progression or death from any cause.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental
Number analyzed (Participants) | 13
months | 5.45 [1.25 to 7.82]

4. Secondary Outcome: Overall Survival (OS)
Description: overall survival (OS) of subjects from the time of enrollment to death from any cause.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental
Number analyzed (Participants) | 13
months | 7.21 [4.5 to 13.77]

5. Secondary Outcome: Safety and Tolerability
Description: Number of participants with a treatment-related adverse events as assessed by an Investigator according to CTCAE v4.0
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 13
Participants | 11

ADVERSE EVENTS:
Time Frame: All AEs from the time of treatment through 30 days following cessation of study treatment and all AEs meeting serious criteria, from the time of treatment through 90 days following cessation of study treatment, or 30 days following cessation of study treatment if the participant initiates new anticancer therapy, whichever is earlier. Up to 2.5 years. All-Cause Mortality monitored up to 3 years.
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 10/14
Serious Adverse Events (participants affected / at risk) | 5/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=14)
Blood bilirubin increased (Investigations) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) — Mental status change
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=14)
Anemia (Blood and lymphatic system disorders) | 7 (9)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (5)
Fever (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Hepatic infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Covid-19
Papulopustular rash (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (3)
Creatinine increased (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (5)
Platelet count decreased (Investigations) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT04306367/Prot_SAP_000.pdf